CLINICAL TRIAL: NCT03609034
Title: Assessment of Knowledge, Attitude and Practice of a Group of Egyptian Dental Interns Toward Caries Risk Assessment and Management:A Cross Sectional Study
Brief Title: Knowledge, Attitude and Practice of a Group of Egyptian Dental Interns Toward Caries Risk Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeel Mustafa Mahmoud El-refaey, Dentist, Cairo University
Other Study IDs: CEBD-CU-2018-06-37
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scientific background(Statement of the problem):

Dental caries is a disease that occurs through complex interaction of four major factors: the host, acidogenic bacteria, fermentable carbohydrates and time. There are many factors which contribute to dental caries incidence but do not seen in clinical examination. Those things are considered as dental caries risk factors, such as socioeconomic, attitudes, knowledge and behavior toward oral health. These risk factors play an important role in incidence of the disease, significantly associated with disease progression . The traditional "drill and fill "concept has served to restore function and esthetics but it has failed to prevent development of new carious lesions. In recent years; better understanding of nature of carious process has changed this operative treatment concept to non destructive risk -based caries management. Caries risk assessment is a procedure used to predict dental caries development before clinical onset of disease, through assessing risk factors contributing to progress of dental caries and let oral health care professionals to be more active in identifying and referring high risk patients for proper treatment and required prevention.

Rationale for carrying out this study : Many studies have measured dentists' knowledge toward caries risk assessment all over the world, but no studies have examined Egyptian Dentists' subjective ratings of the importance of specific caries risk factors or tested whether they use this information in treatment planning.

So the aim of this study to assess knowledge, attitude and practice toward caries risk assessment and management among group of dental interns in Egypt.

Benefits to the Dental interns:

* Challenge the knowledge of the intern dentists regarding caries risk assessment.
* Encourage the concept of minimally invasive dentistry to be applied in clinical practice.
* Accurate caries risk assessment in patients can guide clinician to give attention of their resources to high risk patients.

Benefits to the patients:

* Will benefit from proper knowledge, attitude and practice of dentists, thus proper treatment will be provided.
* Behavioral modification of patients toward oral hygiene practices.
* Reducing patient risk of developing advanced disease and may even arrest disease process.

Benefits to the Community:

-Imparting knowledge of Caries risk assessment to dentists will benefit their patients especially high-caries risk patients by giving proper preventive interventions that help to reduce the expected elevated incidence and severity of caries in the future, therefore the whole community will benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian dental interns who completed their Pediatric Dentistry round in Pediatric Dentistry and Public Health Department ,Faculty of Dentistry , Cairo University.
2. Intern dentists irrespective of age and sex.

Exclusion Criteria:

1. Undergraduate dental students.
2. Post graduate dentists.
3. Dental interns who refused to participate in the study.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All Egyptian dental interns that completed their Pediatric Dentistry round in Pediatric and Dental Public Health Department ,Faculty of Dentistry ,Cairo University during 1 year period.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
knowledge,attitude and practice of dental interns toward caries risk assessment | one year
  structured self-administrated questionnaire

IPD SHARING:
Plan to Share IPD: Undecided